CLINICAL TRIAL: NCT04708119
Title: Histopathologic Changes in Dental Follicle Associated With Radiographically Normal Impacted Lower Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ahmet Altan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-KAEK-081
Record Dates: First submitted 2021-01-06; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Follicle Cyst; Teeth, Impacted; Pathology
MeSH Terms: conditions — Follicular Cyst; Tooth, Impacted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- histopathological evaluation (Other): angulation of impacted lower mandibular third molar and histopathological evaluation
  Interventions: Procedure: The follicular tissues were also excised after tooth extraction.

INTERVENTIONS:
Procedure: The follicular tissues were also excised after tooth extraction. — The follicular tissues were also excised after tooth extraction. Soft tissue samples taken during surgical removal of ILTM were evaluated in the department of pathology.

SUMMARY:
This study aimed to evaluate the incidence of histopathologic changes in dental follicles associated with radiographically normal impacted lower third molar and to determine the relationship between cystic changes in follicle tissues and age, gender, and the angular position of the impacted tooth.

DETAILED DESCRIPTION:
Patients One hundred one healthy patients whose ILTM were extracted for various reasons in Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery were included in the study. All participants included in the study signed an informed consent form. The study was conducted in accordance with the Declaration of Helsinki, and the protocol was approved by Tokat Gaziosmanpaşa University Clinical Research Ethics Committee for the study (Project number: 19-KAEK-081).

The patients' panoramic radiographs were examined, and the impacted teeth were divided into four groups as vertical, horizontal, mesioangular, and distoangular according to their angular positions. The radiographically found that patients with a follicular width of less than 2.5 mm were included in the study. The follicular tissues were also excised after tooth extraction. Soft tissue samples taken during surgical removal of ILTM were evaluated in the department of pathology.

Histopathological evaluation The excision materials obtained for the study were subjected to routine tissue follow-up procedures in Tokat Gaziosmanpaşa University, Faculty of Medicine, Pathology Department. The samples were fixed in 10% formalin solution for 24 hours for light microscope examination and blocked using the routine paraffin blocking method. The preparations were prepared by obtaining sections with microtome from the blocks. These preparations were stained with Hematoxylin Eosin and evaluated under a light microscope. In the histopathological examination, squamous epithelium, keratinization, odontogenic epithelial residue, and fibrosis were evaluated as either present or absent, and inflammation was scored as 0-absent, 1-mild, 2-moderate, or 3-severe. During the microscopic evaluation of follicular tissues, soft tissue samples with stratified squamous epithelium were identified as cystic.

The relationship between histopathological changes observed in the radiographically normal dental follicles and gender and the teeth' angular positions was statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

The radiographically found that patients with a follicular width of less than 2.5 mm were included in the study

Exclusion Criteria:

individuals with systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Data collection | data collection for the first three months,
  The follicular tissues were also excised after tooth extraction
Histopathological examination | histopathological examination for 3 months
  The excision materials obtained for the study were subjected to routine tissue follow-up procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmet Altan, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided